CLINICAL TRIAL: NCT05471960
Title: Neuroplasticity in REM Sleep Behavior Disorder
Brief Title: Neuroplasticity in RBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NEUR-2022-30985
Record Dates: First submitted 2022-07-20; First posted 2022-07-25 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: REM Sleep Behavior Disorder
Keywords: iRBD
MeSH Terms: conditions — REM Sleep Behavior Disorder

STUDY DESIGN:
Intervention Model Description: Prospective (assessments at baseline and 24 months) cross sectional design. Two groups (iRBD, controls)
Masking Description: Outcome assessor will be blind to the group status during data processing and analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iRBD Group: Progression over time (Other): Each subject be assessed at baseline and approximately 2 years later. At each time point, each participant will attend eight testing sessions (MRI scanning, two TMS-motor test visits, two TMS-prefrontal test visits, motor assessments, neuropsychological testing, and overnight sleep testing (polysomnography - PSG).
  Interventions: Other: Natural progression over time
- Control Group: Progression over time (Other): Each subject be assessed at baseline and approximately 2 years later. At each time point, each participant will attend eight testing sessions (MRI scanning, two TMS-motor test visits, two TMS-prefrontal test visits, motor assessments, neuropsychological testing, and overnight sleep testing (polysomnography - PSG).
  Interventions: Other: Natural progression over time

INTERVENTIONS:
Other: Natural progression over time — Each subject will attend eight testing sessions (MRI scanning, two TMS-motor test visits, two TMS-prefrontal test visits, motor assessments, neuropsychological testing, and overnight sleep testing (polysomnography - PSG).

SUMMARY:
REM sleep behavior disorder is a parasomnia that reflects the presence of alpha-synucleinopathy in the brain and is highly predictive of eventual phenoconversion to Parkinson's disease, dementia with Lewy bodies, or multiple system atrophy over the course of years to decades. Neuroplastic adaptations in the brain during the prodromal stage of disease are thought to mask the expression of motor and non-motor signs and may substantially delay diagnosis during a potentially critical time window. This study will examine the state and progression (over 30 to 36 months) of neuroplastic changes in the excitability of the motor and prefrontal cortex (using transcranial magnetic stimulation), the structural and functional connectivity of the brain (using highfield, 7T, magnetic resonance imaging), and the relationship of these changes to the expression of motor and neuropsychological signs, in a cohort of individuals with REM sleep behavior disorder and matched controls.

ELIGIBILITY:
Inclusion Criteria for the iRBD Group:

* Diagnosis of polysomnogram-confirmed isolated iRBD.
* Able to ambulate independently without the use of an assistive device (e.g., cane) for 50 meters.
* Age: 21-75 years.

Inclusion Criteria For Control Subject Group:

* Age: 21-75 years.
* Able to ambulate independently without the use of an assistive device (e.g., cane or walker for 50 meters.

Exclusion criteria for iRBD group:

* Dementia diagnosis and/or a University of California Brief Assessment of Capacity to Consent (UBACC) score and MacCAT-CR score indicating impaired capacity to consent.
* History of musculoskeletal disorders that significant affect movement of lower or upper limbs as determined at the time of enrollment.
* Other significant neurological disorders that may affect participation or performance in the study.
* Anti-depressant associated RBD. Individuals will be excluded if their dream enactment emerged or clearly worsened after initiating an antidepressant medication.
* Meet criteria for overt Parkinson's disease, dementia with Lewy bodies, Multiple Systems Atrophy, Alzheimer's disease, or other neurodegenerative disorder, or other known cause of RBD (e.g., narcolepsy and drug induced RBD).
* Untreated sleep-disordered breathing
* History of musculoskeletal disorders that significantly affect movement of lower or upper limbs as determined at the time of enrollment.
* Pregnant women
* Additional exclusion criteria for TMS experiments (note that individuals who are excluded from the TMS experiment still have the opportunity to participate in the other data collection sessions):

  * History of seizures, epilepsy, stroke, multiple sclerosis, or traumatic brain injury
  * Recent history of frequent syncope (fainting) episodes in response to blood, emotional stress, or sensory triggers.
  * Intracranial metallic or magnetic devices (e.g. cochlear implant, deep brain stimulator)
  * Pacemaker or any implanted device
  * History of surgery on blood vessels, brain, or heart
  * Unexplained, recurring headaches or concussion within the last six months
  * Severe hearing impairment
  * If participant is taking one of the following medications that affects neuroplasticity testing, they will be excluded from the TMS experiment: haloperidol (dopamine antagonist), prazosin (norepinephrine antagonist), biperiden (acetylcholine antagonist), dopamine modulators, NMDA receptor and calcium channel modulators, GABAergic drugs (benzodiazepines), lithium, lovastatin, and cannabis.

Exclusion Criteria for Control subject Group:

* Same as exclusion criteria as the iRBD group
* History of dream enactment from either patient report or from a bed partner witness that may suggest iRBD.
* History of untreated sleep-disordered breathing.
* Presence of parkinsonism or cognitive impairment (including dementia or mild cognitive impairment).
* Active central nervous system, systemic, psychiatric conditions or use of psychoactive medication that would adversely affect cognitive, neuropsychiatric, motor, or autonomic functioning

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2030-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
MRI Progression over 30 to 36 months | 30 to 36 months from baseline
  Yes/No whether a change was observed from baseline
Change in Beck Depression Inventory score | 30 to 36 months from baseline
  Higher score means more impairment
Change in Mattis Dementia Rating Scale | 30 to 36 months from baseline
  Higher score means less impairment
Change in Rey Complex Figure | 30 to 36 months from baseline
  Higher score means less impairment
Change in WAIS-IV Matrix Reasoning | 30 to 36 months from baseline
  Higher score means less impairment
Change in Stroop Color | 30 to 36 months from baseline
  Higher score means less impairment
Change in Stroop Word | 30 to 36 months from baseline
  Higher score means less impairment
Change in Stroop Color Word | 30 to 36 months from baseline
  Higher score means less impairment
Change in Wisconsin Card Sorting Test | 30 to 36 months from baseline
  Higher score means more impairment for subsections "# persev errors" and FMS; less impairment for subsections "# categories" and conceptualization
Change in D-KEFS | 30 to 36 months from baseline
  Higher score means less impairment
Change in BVMT-R | 30 to 36 months from baseline
  Higher score means less impairment
Change in HVLT | 30 to 36 months from baseline
  Higher score means less impairment
Change in WMS-3 Spatial Span | 30 to 36 months from baseline
  Higher score means less impairment
Change in Boston Naming Test | 30 to 36 months from baseline
  Higher score means less impairment
Change in Trail Making Test A | 30 to 36 months from baseline
  Higher score means more impairment
Change in Trail Making Test B | 30 to 36 months from baseline
  Higher score means more impairment

CONTACTS AND LOCATIONS:
Overall Officials: Colum MacKinnon, Ph.D, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States